CLINICAL TRIAL: NCT04872959
Title: TRANSFORM Heart Failure with Reduced Ejection Fraction
Acronym: TRANSFORMHFrEF
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: sponsor decision
Sponsor: Massachusetts General Hospital (Other)
Collaborators: American College of Cardiology (Other)
Responsible Party: Principal Investigator, James L. Januzzi, Principal Investigator, Massachusetts General Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Pro00047392
Record Dates: First submitted 2021-04-26; First posted 2021-05-05 (Actual); Last update posted 2024-11-20 (Actual); Status verified 2024-11

CONDITIONS: Heart Failure, Systolic
MeSH Terms: conditions — Heart Failure, Systolic

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Usual Care Arm (No Intervention): Will not use HealthReveal to titrate the doses of Entresto/ other treatments for HFrEF.
- Interventional- Health Reveal (Experimental): The interventional arm will be provided tools to augment quality of care and build the patient and physician relationship through trust and shared goal-setting.
  Prior to each patient appointment, on a customized GDMT Dashboard, the site will receive a pre-visit assessment of GDMT accompanied by recommended adjustment(s) using information extracted weekly from the sites' electronic health record (EHR). The recommended adjustment(s) will be conveyed using proprietary software from HealthReveal, with a suggested follow up plan. All reminders regarding dosing targets are based on the 2020 ACC Expert Consensus Decision Pathway for Optimization of Heart Failure Treatment.
  Additionally, during visits at baseline, 3 months, and 6 months, patient-reported outcomes/QOL will be assessed.
  Interventions: Other: HealthReveal

INTERVENTIONS:
Other: HealthReveal — In the Intervention arm, for each study visit, the site will receive a pre-visit assessment of GDMT accompanied by recommended adjustment(s) using information extracted weekly from the sites' EHR.
  The recommended adjustment(s) will be conveyed using proprietary software from HealthReveal, with a suggested follow up plan. All reminders regarding dosing targets are based on the 2020 ACC Expert Consensus Decision Pathway for Optimization of Heart Failure Treatment.
  Additionally, during visits at baseline, 3 months, and 6 months, the KCCQ-23 will be completed.
  In the Usual Care arm, during visits at baseline, 3 months, and 6 months, the KCCQ-23 will be completed.
  Arms: Interventional- Health Reveal

SUMMARY:
The goal of the TRANSFORM-HFrEF trial will be to study the current guideline-directed medical therapy (GDMT) landscape for HFrEF and determine effective methods and models of increasing adherence to GDMT and improving Quality of Life (QOL) in outpatient settings within the context of the 20-minute visit. This will be achieved through a randomized evaluation that shifts standard clinical interview and documentation requirements outside the office visit and building the patient and physician relationship through trust and shared goal setting.

Specific Aims:

To evaluate the ability of ACC Solution Sets and Patient Resources to improve initiation and titration of GDMT for eligible patients with HFrEF Left Ventricle Ejection Fraction (LVEF) ≤ 40%.

To evaluate change in QOL between patients in the intervention arm and the Usual Care arm.

Examine the relative change in GDMT among higher risk versus lower-risk patients in the Intervention arm and Usual Care arm.

In this randomized registry trial, sites will be invited to participate in a 6-month study aimed at various processes of care in HFrEF. Sites would be informed that they might be asked to participate in an intensive intervention to improve GDMT prescription or in a study of QOL in HFrEF. Once a list of sites interested in participating is created, sites would be randomized into two arms: an intervention group and a usual care group.

DETAILED DESCRIPTION:
Heart Failure (HF) is the cardiovascular epidemic of the 21st century, affecting millions of patients worldwide. It is believed that HF is the only cardiovascular diagnosis rising in incidence among elderly patients and is the #1 diagnosis leading to hospitalization among Medicare recipients. In addition to being increasingly prevalent, HF has a poor outlook after initial diagnosis and is associated with poor quality of life (QOL) in affected patients; this not only leads to the burden on patients, family, and other caregivers but also on the healthcare system. For all these reasons, optimizing the understanding and care of patients with HF is a major priority.

Although clinical practice guidelines clearly articulate optimal GDMT for the care of patients with HFrEF, implementation of GDMT into the management of such patients has proven to be suboptimal, with most patients under-treated relative to goal therapy.

To evaluate the contemporary status of GDMT delivery for HFrEF, the recent Change the Management of Patients with Heart Failure (CHAMP-HF) registry included 3518 patients from 150 primary care and cardiology practices (1,2). The mean age of this cohort was 66 ± 13 years, 29% were female, and mean EF was 29 ± 8%, thus representing a very characteristic population of patients with HFrEF.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years
* Clinical diagnosis of HF with EF ≤40% documented within 1 year of enrollment
* Receiving ≥1 oral medication for HF at study enrollment (including diuretics, ACEI/ARB/ARNI, beta-blockers, MRA, SGLT2i or thiazide diuretics.

Exclusion Criteria:

* Current or anticipated participation in a clinical trial
* Currently receiving comfort care or enrolled in hospice
* Life expectancy <1 year
* History of or plan for heart transplantation or left ventricular assist device
* Current or planned hemodialysis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2021-10-22 (Actual); Primary Completion 2023-01-01 (Actual); Study Completion 2024-05 (Estimated)

PRIMARY OUTCOMES:
average composite endpoint of target dose achievement for the main classes of drugs (RASi/beta blockers/MRA/SGLT2i) among eligible patients without documented contraindications or intolerance. | baseline to 6 months
  From baseline to 6 months change in average composite endpoint of target dose achievement for the main classes of drugs (RASi/beta blockers/MRA/SGLT2i) among eligible patients without documented contraindications or intolerance. Goal doses will be based on the 2020 ACC Expert Consensus Decision Pathway for Optimization of Heart Failure Treatment (4).
  Numerator = receiving ARNI/ACEI/ARB at 50% or higher of target dose + receiving evidence-based beta blocker at 50% or higher of target dose + receiving MRA at 50% or higher of target dose + receiving SGLT2i at 50% or higher of target dose.
  Denominator = eligible to receive ARNI/ACEI/ARB and no documented reason for not receiving higher dose, eligible to receive evidence-based beta blocker and no documented reason for not receiving higher dose.

SECONDARY OUTCOMES:
Relative change in actual achieved doses of individual classes of pivotal therapies (RASi/beta blocker/ MRA/SGLT2i). | baseline to 6 months
  1) Relative change in actual achieved doses of individual classes of pivotal therapies (RASi/beta blocker/ MRA/SGLT2i).
change in achievement of target doses | baseline to 6 months
  2) Relative change in achievement of target doses (yes/no) of pivotal therapies (RASi/beta blocker/MRA/SGLT2i).

IPD SHARING:
Plan to Share IPD: Undecided
results

REFERENCES:
- [Background] DeVore AD, Thomas L, Albert NM, Butler J, Hernandez AF, Patterson JH, Spertus JA, Williams FB, Turner SJ, Chan WW, Duffy CI, McCague K, Mi X, Fonarow GC. Change the management of patients with heart failure: Rationale and design of the CHAMP-HF registry. Am Heart J. 2017 Jul;189:177-183. doi: 10.1016/j.ahj.2017.04.010. Epub 2017 Apr 29. PMID 28625374
- [Background] Greene SJ, Butler J, Albert NM, DeVore AD, Sharma PP, Duffy CI, Hill CL, McCague K, Mi X, Patterson JH, Spertus JA, Thomas L, Williams FB, Hernandez AF, Fonarow GC. Medical Therapy for Heart Failure With Reduced Ejection Fraction: The CHAMP-HF Registry. J Am Coll Cardiol. 2018 Jul 24;72(4):351-366. doi: 10.1016/j.jacc.2018.04.070. PMID 30025570
- [Background] Ibrahim NE, Song Y, Cannon CP, Doros G, Trebnick A, Russo P, Ponirakis A, Alexanian C, Januzzi JL Jr. Retraction notice to Addition or removal of guideline directed medical therapy in ambulatory patients with heart failure with reduced ejection fraction relative to change in symptom severity: An analysis from the PINNACLE (Practice Innovation and Clinical Excellence) Registry(R) [International Journal of Cardiology 254 (2018) 222-223]. Int J Cardiol. 2018 Mar 1;254:R1. doi: 10.1016/j.ijcard.2018.05.008. No abstract available. PMID 29752128
- [Background] Yancy CW, Januzzi JL Jr, Allen LA, Butler J, Davis LL, Fonarow GC, Ibrahim NE, Jessup M, Lindenfeld J, Maddox TM, Masoudi FA, Motiwala SR, Patterson JH, Walsh MN, Wasserman A. 2017 ACC Expert Consensus Decision Pathway for Optimization of Heart Failure Treatment: Answers to 10 Pivotal Issues About Heart Failure With Reduced Ejection Fraction: A Report of the American College of Cardiology Task Force on Expert Consensus Decision Pathways. J Am Coll Cardiol. 2018 Jan 16;71(2):201-230. doi: 10.1016/j.jacc.2017.11.025. Epub 2017 Dec 22. No abstract available. PMID 29277252